CLINICAL TRIAL: NCT01191060
Title: Randomized Study Comparing Conventional Dose Treatment Using a Combination of Lenalidomide, Bortezomib and Dexamethasone to High-Dose Treatment With ASCT in the Initial Management of Myeloma in Patients up to 65 Years of Age
Brief Title: Study Comparing Conventional Dose Combination RVD to High-Dose Treatment With ASCT in the Initial Myeloma up to 65 Years
Acronym: IFM/DFCI2009
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Celgene Corporation (Industry); Janssen-Cilag Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09 110 01
Record Dates: First submitted 2010-04-16; First posted 2010-08-30 (Estimated); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Myeloma
Keywords: Progression free survival prolongation; Disease Progression; Overall survival
MeSH Terms: conditions — Neoplasms, Plasma Cell; Disease Progression | interventions — Lenalidomide; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- lenalidomide, bortezomib with ASCT (Experimental): RVD q 21 days (2 cycles) Collection of peripheral blood stem cells (PBSCs) using cyclophosphamide and GCSF (type Granocyte® or equivalent)
  Autologous stem cell transplant:
  Melphalan: infused over two days (day -2 and day -1) or as a single infusion (day-2) according to institutional practice Re-infusion of PBSCs RVD q 21 days (2 cycles) Maintenance Lenalidomide q28 days (12 months)
  Interventions: Drug: Lenalidomide, Bortezomib
- lenalidomide, bortezomib without ASCT (Experimental): RVD q 21 days (2 cycles) Collection of peripheral blood stem cells (PBSCs) using cyclophosphamide and GCSF (type Granocyte® or equivalent) RVD q 21 days (5 cycles) Maintenance Lenalidomide q28 days (12 months)
  Interventions: Drug: Lenalidomide, Bortezomib

INTERVENTIONS:
Drug: Lenalidomide, Bortezomib — Lenalidomide/Bortézomib/Dexamethasone cycles:
  Number of cycles: 8 cycles for arm A
  Cycle length
  Dosage:
  * Lenalidomide: 25 mg/day on days 1-14 of each cycle
  * Bortézomib: 1.3 mg/m2 on days 1, 4, 8, and 11 for 1 cycle of each cycle
  Maintenance phase (12 months):
  Cycle length: 28 days Dosage: Lenalidomide: 10 mg/day continuously for 28 days during 3 months and if the participant tolerates 10 mg/day without complication, a dose increase to 15 mg/day will be allowed
  Other Names: Lenalidomide (REVLIMID®); Bortezomib (VELCADE®)
  Arms: lenalidomide, bortezomib without ASCT
Drug: Lenalidomide, Bortezomib — Lenalidomide Bortezomib Dexamethasone cycles:
  Number of cycles: 5 cycles for arm B
  Cycle length
  Dosage:
  * Lenalidomide: 25 mg/day on days 1-14 of each cycle
  * Bortézomib: 1.3 mg/m2 on days 1, 4, 8, and 11 for 1 cycle of each cycle
  Maintenance phase (12 months):
  Cycle length: 28 days Dosage: Lenalidomide: 10 mg/day continuously for 28 days during 3 months and if the participant tolerates 10 mg/day without complication, a dose increase to 15 mg/day will be allowed
  Other Names: Lenalidomide (REVLIMID®); Bortézomib (VELCADE®)
  Arms: lenalidomide, bortezomib with ASCT

SUMMARY:
Objective of this study is to determine if, in the era of novel drugs, high dose therapy (HDT) is still necessary in the initial management of multiple myeloma in younger patients. HDT as compared to conventional dose treatment would be considered superior if it significantly prolongs Progression-free survival (by at least 9 months).

DETAILED DESCRIPTION:
Study design Phase III, multicenter, randomized, open-label study designed to evaluate the clinical benefit from the drug combination RVD without immediate high-dose therapy (HDT) followed by lenalidomide maintenance (Arm A) versus RVD plus HDT and PBSCT followed by lenalidomide maintenance (Arm B).

ELIGIBILITY:
Inclusion Criteria for registration :

(with labs performed within 21 days of initiation of protocol therapy):

* Patients diagnosed with multiple myeloma based on International Myeloma Foundation 2003 Diagnostic Criteria.
* Patients must have symptomatic myeloma with myeloma-related organ damage.
* Patients must have myeloma that is measurable by either serum or urine evaluation of the monoclonal component or by assay of serum free light chains.
* Age between 18 and 65 years at the time of signing the informed consent document.
* ECOG performance status <2 (Karnofsky ≥ 60%)
* Negative HIV blood test

Exclusion Criteria for registration (section 4.2):

* Participants must not have been treated with any prior systemic therapy for multiple myeloma. Treatment by localized radiotherapy is not an exclusion criterion if an interval of at least two weeks between the end of radiotherapy and initiation of protocol therapy entry in the study is observed. Similarly, the dose of corticosteroids received by the participant should not exceed the equivalent of 160 mg of dexamethasone over a two-week period before initiation of protocol therapy.
* Primary amyloidosis (AL) or myeloma complicated by amylosis.
* Participants may not be receiving any other study investigational agents.
* Participants with known brain metastases
* Poor tolerability or known allergy to any of the study drugs or compounds of similar chemical or biologic composition to study agents
* Platelet count < 50,000/mm3 per µLwithin 21 days of initiation of protocol therapy. Transfusion within 7 days of screening is not allowed to meet platelet eligibility criteria.
* ANC < 1,000 cells/mm3 within 21 days of initiation of protocol therapy. Growth factor within 7 days of screening is not allowed to meet ANC eligibility criteria.
* Hemoglobin < 8.0 g/dL within 21 days of initiation of protocol therapy. Transfusion may be used to meet hemoglobin eligibility criteria.
* Hepatic impairment, defined a bilirubin > 1.5 x institutional upper limit of normal (ULN) > 2 mg/dL (Patients with benign hyperbilirubinemia (e.g., Gilbert's syndrome) are eligible) and or AST (SGOT), or ALT (SGPT), or alkaline phosphatase > 2 x ULN
* Renal insufficiency, defined as serum creatinine > 2.5 mg/dl and/or creatinine clearance < <40 60 ml/min (actual or calculated). The Cockgroft-Gault formula should be used for calculating creatinine clearance values, and may be located in Section 4.2
* Respiratory compromise, defined as ventilation tests and with DLCO < 50%
* Participant must not demonstrate with clinical signs of heart or coronary failure, or evidence of LVEF < 40%. Participant must not have with myocardial infarction within 6 months prior to enrollment or have New York Heart Association (NYHA Appendix VII) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at screening has to be documented by the investigator as not medically relevant.
* Intercurrent illness including, but not limited to ongoing or active severe infection, known (active or not) infection with hepatitis B or C virus, poorly controlled diabetes, severe uncontrolled psychiatric disorder or psychiatric illness/social situations that would limit compliance with study requirements.
* Participant with previous history of another malignant condition, except for basal cell carcinoma and stage I cervical cancer
* Female participant who is pregnant or breast-feeding
* Inability to comply with an anti-thrombotic treatment regimen
* Peripheral neuropathy ≥ Grade 2 peripheral neuropathy on clinical examination within 21 days of initiation of protocol therapy
* Mental illness likely to interfere with participation in the study and Adults under juridical protection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Actual)
Dates: Start 2010-10 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival | up to 4 years
  To compare progression-free survival (PFS) between the Arm A and Arm B up to 4 years or until progression

SECONDARY OUTCOMES:
Response Rates | up to 4 years
  -Response rates (RR) between the two arms up to 4 years or until progression
Time To Progression | up to 4 years
  Time to progression (TTP) between the two arms up to 4 years or until progression
Toxicity comparison | up to 4 years
  Toxicity comparison between the two arms randomization up to 4 years or until progression
Genetic prognostic groups definition | up to 4 years
  Genetic prognostic groups definition (evaluated by gene expression profiling-GEP) from randomization up to 4 years or until progression
Best treatment examination in each GEP-defined prognostic group. | up to 4 years
  Best treatment examination in each GEP-defined prognostic group. from randomization up to 4 years or until progression

CONTACTS AND LOCATIONS:
Overall Officials: MICHEL ATTAL, MD PhD, Principal Investigator — University Hospital of Toulouse
Locations (68):
- France (68):
  - CH du Pays D'Aix, Aix-en-Provence
  - CHRU - Hôpital Sud Amiens, Amiens
  - CHU d'Angers, Angers
  - Centre Hospitalier Argenteuil Victor Dupouy, Argenteuil
  - Centre Hospitalier H.Duffaut, Avignon
  - Centre Hospitalier de la côte basque, Bayonne
  - Hôpital Jean Minjoz, Besançon
  - Centre Hospitalier de Blois, Blois
  - Hôpital Avicenne, Bobigny
  - Polyclinique Bordeaux Nord Aquitaine, Bordeaux
  - Hôpital A.Morvan, Brest
  - CHU Caen Côte de Nacre, Caen
  - Centre François Baclesse, Caen
  - CH René Dubos, Cergy-Pontoise
  - Centre Hospitalier William Morey, Chalon-sur-Saône
  - CH Chambéry, Chambéry
  - Hôpital Antoine Béclère, Clamart
  - Hôpital d'instruction des armées Percy, Clamart
  - CHU d'Estaing, Clermont-Ferrand
  - Pole Santé République, Clermont-Ferrand
  - CH Louis Pasteur - Colmar, Colmar
  - CH Sud Francilien, Corbeil-Essonnes
  - CHU Henri Mondor, Créteil
  - CHRU Dijon, Dijon
  - Centre Hospitalier Général - Dunkerque, Dunkirk
  - Hôpital A.Michallon, Grenoble
  - Centre hospitalier départemental - La Roche sur Yon cedex, La Roche-sur-Yon
  - CH de Chartres - Hôpital Louis Pasteur, Le Coudray
  - Centre Jean Bernard, Le Mans
  - Centre hospitalier Le Mans, Le Mans
  - CHRU - Hôpital Claude Huriez, Lille
  - CHU de Limoges, Limoges
  - Centre hospitalier Bodelio, Lorient
  - CHU - Hôpital Edouard Herriot, Lyon
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmettes, Marseille
  - CH Meaux, Meaux
  - Hopital E Muller, Mulhouse
  - Hôpitaux de Brabois, Nancy
  - Centre Catherine de Sienne, Nantes
  - CHRU - Hôtel Dieu, Nantes
  - Hôpital Archet 1, Nice
  - Hôpital de l'Archet, Nice
  - Groupe Hospitalo-Universitaire Carémeau, Nîmes Cédex 9
  - Institut Curie, Paris
  - Hôpital Cochin, Paris
  - Hôpital Saint-Louis, Paris
  - Hôpital St-Antoine, Paris
  - CH Saint Jean, Perpignan
  - CHRU - Hôpital du Haut Lévêque, Pessac
  - Centre Hospitalier Lyon sud, Pierre-Bénite
  - CHRU - Hôpital Jean Bernard, Poitiers
  - Centre Hospitalier de la région d'Annecy, Pringy
  - Hôpital R.Debré, Reims
  - CHRU - Hôpital de Pontchaillou, Rennes
  - CHRU - Hôpital Sud, Rennes
  - Centre Henri Becquerel, Rouen
  - Centre Hospitalier Yves le Foll, Saint-Brieuc
  - Centre René Huguenin, Saint-Cloud
  - Centre Hospitalier Départemental - La réunion St Denis, Saint-Denis
  - Groupe Hospitalier Sud Réunion, Saint-Pierre
  - Institut de Cancérologie de la Loire, Saint-Priest-en-Jarez
  - Hôpitaux Universitaires de Strasbourg, Strasbourg
  - University Hospital of Toulouse, Purpan, Toulouse
  - CHRU - Hôpital Bretonneau, Tours
  - Centre Hospitalier de Valence, Valence
  - CH Bretagne Atlantique Vannes et Auray, Vannes
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Derived] Rosinol L, Hebraud B, Oriol A, Colin AL, Rios Tamayo R, Hulin C, Blanchard MJ, Caillot D, Sureda A, Hernandez MT, Arnulf B, Mateos MV, Macro M, San-Miguel J, Belhadj K, Lahuerta JJ, Garelik MB, Blade J, Moreau P. Integrated analysis of randomized controlled trials evaluating bortezomib + lenalidomide + dexamethasone or bortezomib + thalidomide + dexamethasone induction in transplant-eligible newly diagnosed multiple myeloma. Front Oncol. 2023 Nov 2;13:1197340. doi: 10.3389/fonc.2023.1197340. eCollection 2023. PMID 38023148
- [Derived] Noori S, Wijnands C, Langerhorst P, Bonifay V, Stingl C, Touzeau C, Corre J, Perrot A, Moreau P, Caillon H, Luider TM, Dejoie T, Jacobs JFM, van Duijn MM. Dynamic monitoring of myeloma minimal residual disease with targeted mass spectrometry. Blood Cancer J. 2023 Feb 24;13(1):30. doi: 10.1038/s41408-023-00803-z. No abstract available. PMID 36828828
- [Derived] Langerhorst P, Noori S, Zajec M, De Rijke YB, Gloerich J, van Gool AJ, Caillon H, Joosten I, Luider TM, Corre J, VanDuijn MM, Dejoie T, Jacobs JFM. Multiple Myeloma Minimal Residual Disease Detection: Targeted Mass Spectrometry in Blood vs Next-Generation Sequencing in Bone Marrow. Clin Chem. 2021 Nov 26;67(12):1689-1698. doi: 10.1093/clinchem/hvab187. PMID 34643690
- [Derived] Samur MK, Aktas Samur A, Fulciniti M, Szalat R, Han T, Shammas M, Richardson P, Magrangeas F, Minvielle S, Corre J, Moreau P, Thakurta A, Anderson KC, Parmigiani G, Avet-Loiseau H, Munshi NC. Genome-Wide Somatic Alterations in Multiple Myeloma Reveal a Superior Outcome Group. J Clin Oncol. 2020 Sep 20;38(27):3107-3118. doi: 10.1200/JCO.20.00461. Epub 2020 Jul 20. PMID 32687451
- [Derived] Roussel M, Hebraud B, Hulin C, Perrot A, Caillot D, Stoppa AM, Macro M, Escoffre M, Arnulf B, Belhadj K, Karlin L, Garderet L, Facon T, Guo S, Weng J, Dhanasiri S, Leleu X, Moreau P, Attal M. Health-related quality of life results from the IFM 2009 trial: treatment with lenalidomide, bortezomib, and dexamethasone in transplant-eligible patients with newly diagnosed multiple myeloma. Leuk Lymphoma. 2020 Jun;61(6):1323-1333. doi: 10.1080/10428194.2020.1719091. Epub 2020 Feb 22. PMID 32090636
- [Derived] Attal M, Lauwers-Cances V, Hulin C, Leleu X, Caillot D, Escoffre M, Arnulf B, Macro M, Belhadj K, Garderet L, Roussel M, Payen C, Mathiot C, Fermand JP, Meuleman N, Rollet S, Maglio ME, Zeytoonjian AA, Weller EA, Munshi N, Anderson KC, Richardson PG, Facon T, Avet-Loiseau H, Harousseau JL, Moreau P; IFM 2009 Study. Lenalidomide, Bortezomib, and Dexamethasone with Transplantation for Myeloma. N Engl J Med. 2017 Apr 6;376(14):1311-1320. doi: 10.1056/NEJMoa1611750. PMID 28379796
- [Derived] Dunavin NC, Wei L, Elder P, Phillips GS, Benson DM Jr, Hofmeister CC, Penza S, Greenfield C, Rose KS, Rieser G, Merritt L, Ketcham J, Heerema N, Byrd JC, Devine SM, Efebera YA. Early versus delayed autologous stem cell transplant in patients receiving novel therapies for multiple myeloma. Leuk Lymphoma. 2013 Aug;54(8):1658-64. doi: 10.3109/10428194.2012.751528. Epub 2012 Dec 31. PMID 23194056